CLINICAL TRIAL: NCT00000628
Title: A Pharmacokinetic Study of L-697,661 Alone and in Combination With Zidovudine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 184; Merck Protocol 020-00
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 1994-10

CONDITIONS: HIV Infections
Keywords: Drug Evaluation; Drugs, Investigational; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Drug: L-697,661
Drug: Zidovudine

SUMMARY:
Part 1: To study the potential safety and pharmacokinetic (blood level) effects of zidovudine (AZT) on L-697,661; to obtain additional pharmacokinetic information in humans with L-697,661; to study the effect of L-697,661 on hepatic enzyme induction. Part 2: To begin a study of the antiviral activity of L-697,661.

L-697,661 is a newly identified compound that inhibits HIV replication (reproduction and growth) in cell culture. It works together with AZT against HIV.

DETAILED DESCRIPTION:
L-697,661 is a newly identified compound that inhibits HIV replication (reproduction and growth) in cell culture. It works together with AZT against HIV.

Part 1: Twelve patients are randomly assigned to one of two groups. Group 1 patients receive AZT for 7 days, followed by AZT plus L-697,661 with food for 56 days. Group 2 patients receive no drug for 7 days, followed by L-697,661 with food for 56 days. Antipyrine is administered 1 hour prior to study drug on days 8, 22, and 35.

Part 2: Fifteen patients receive L-697,661 with food, for 8 weeks. Therapy with L-697,661 may be extended beyond 8 weeks for up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.

Prior Medication: Included:

* Patients in Part 1 must have received no previous zidovudine (AZT) or a stable dose of at least 500 mg/day without evidence of toxicity.
* Patients in Part 2 must have received no previous AZT or = or > 300 mg/day for < 6 consecutive weeks within 1 year prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Acute HIV-related opportunistic infection requiring ongoing treatment.
* Diarrhea defined as 3 or more liquid stools/day for one week.
* Wilson's or Gilbert's disease, porphyria, or other chronic or acute hepatic disease.
* Potentially life-threatening allergic reactions to any of the components of zidovudine.
* Acute or chronic medical conditions that in the opinion of the investigator would place patient at risk by participation in this study.

Concurrent Medication:

Excluded:

* Systemic bronchodilators, acetaminophen, aspirin.

Prior Medication:

Excluded:

* Didanosine (ddI) or dideoxycytidine (ddC) within 14 days prior to entry.
* Immune modulators or investigational drugs within 30 days prior to entry.
* Drugs known to induce hepatocellular enzymes, such as phenobarbital, phenytoin, warfarin, ketoconazole, and oral contraceptives, within 30 days prior to entry.

Patients in Part 2 only:

Excluded:

* Zidovudine within 4 weeks prior to receiving first dose of study drug.

Risk Behavior:

Excluded:

* Patients who the investigator feels would not comply with study requirements.

Patients may not have the following prior conditions:

* Acute or chronic medical conditions that in the opinion of the investigator would place patient at risk by participation in this study.
* Potentially life-threatening allergic reactions to any of the components of zidovudine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27

CONTACTS AND LOCATIONS:
Overall Officials: RT Schooley, Study Chair
Locations (5):
- United States (5):
  - San Francisco Gen Hosp, San Francisco, California
  - Univ of Colorado Health Ctr / Denver Gen Hosp, Denver, Colorado
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Kuritzkes DR, Curtis S, Rosandich M, Stein DS, Schooley RT. Delayed emergence of resistance to L-697,661 in patients receiving concomitant zidovudine. The ACTG 184 Study Team. Int Conf AIDS. 1993 Jun 6-11;9(1):467 (abstract no PO-B26-1994)
- [Background] Schooley RT, Campbell TB, Kuritzkes DR, Blaschke T, Stein DS, Rosandich ME, Phair J, Pottage JC, Messari F, Collier A, Kahn J. Phase 1 study of combination therapy with L-697,661 and zidovudine. The ACTG 184 Protocol Team. J Acquir Immune Defic Syndr Hum Retrovirol. 1996 Aug 1;12(4):363-70. doi: 10.1097/00042560-199608010-00006. PMID 8673545
- [Background] Campbell TB, Routh JA, Bakhtiari M, Schooley RT, Kuritzkes DR. Detection of genotypic changes in reverse transcriptase during combination therapy with zidovudine and L-697,661. Detection of genotypic changes in reverse transcriptase during combination therapy with zidovudine and L-697,661. Int Conf AIDS. 1993 Jun 6-11;9(1):239 (abstract no PO-A26-0630)